CLINICAL TRIAL: NCT00846248
Title: Chromium and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H847627262
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Insulin Resistance
Keywords: diabetes; insulin resistance; chromium; healthy volunteers
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Chromium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Chromium picolinate
  Interventions: Dietary Supplement: Chromium
- 2 (Placebo Comparator): 2 sugar pills taken twice daily
  Interventions: Dietary Supplement: Chromium; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Chromium — We will enroll non-obese, non-diabetic subjects with insulin resistance in a 16 week treatment program with 500 μg of chromium picolinate twice daily. Insulin action will be determined by insulin clamp and OGTT using deuterated glucose both before and after treatment. Subjects will be compared to a placebo-treated group.
Dietary Supplement: placebo — We will enroll non-obese, non-diabetic subjects with insulin resistance in a 16 week treatment program with 500 μg of chromium picolinate twice daily. Insulin action will be determined by insulin clamp and OGTT using deuterated glucose both before and after treatment. Subjects will be compared to a placebo-treated group.
  Arms: 2

SUMMARY:
Chromium is an essential nutrient for the maintenance of normal glucose tolerance and its deficiency causes insulin resistance. Chromium administration has also been shown in several studies to lower glucose and insulin levels in patients with type 2 diabetes. Accordingly, we propose to perform a placebo-controlled study of chromium picolinate administration in a cohort of non-obese, non-diabetic, insulin resistant subjects. These subjects will be randomized to 16 weeks of therapy with either 500 mcg twice a day of Chromium or placebo.

DETAILED DESCRIPTION:
Chromium is an essential nutrient for the maintenance of normal glucose tolerance and its deficiency causes insulin resistance. Chromium administration has also been shown in several studies to lower glucose and insulin levels in patients with type 2 diabetes. Moreover, studies in humans, animals and cell culture indicate that chromium enhances insulin signaling. While these studies suggest that chromium administration increases insulin sensitivity, it has not been directly demonstrated that chromium has an effect in well defined insulin resistant subjects independent of hyperglycemia. Accordingly, we propose to perform a placebo-controlled study of chromium picolinate administration in a cohort of non-obese, non-diabetic, insulin resistant subjects. The insulin sensitivity of 80 subjects will be measured by a euglycemic insulin clamp. Approximately 40 insulin resistant subjects will be randomized to 16 weeks of therapy with either 500 ug twice a day of chromium picolinate or placebo. To quantitate the chromium-induced improvements, euglycemic hyperinsulinemic clamps to evaluate insulin sensitivity, OGTT using deuterated glucose to evaluate glycolytic glucose disposal, and muscle biopsies to evaluate insulin signaling pathways, will be performed before and after treatment. We believe these studies will (1) confirm the beneficial effect of chromium on insulin sensitivity; (2) further our understanding of the molecular mechanisms of chromium action; and (3) because these insulin resistant subjects are at risk for the development of type 2 diabetes, the Metabolic Syndrome, and coronary artery disease (CAD), a demonstration of the beneficial effects of chromium on insulin action could ultimately have important public health consequences.

ELIGIBILITY:
Inclusion Criteria:

* Not exercising regularly, healthy, non-diabetic.

Exclusion Criteria:

* Diabetes, heart disease, hepatitis, HIV, impaired glucose tolerance, abnormal liver enzymes, abnormal TSH levels, other abnormal lab values.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 0 months and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Masharani, MD, Principal Investigator — University of California, San Francisco; Martha Nolte, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Masharani U, Gjerde C, McCoy S, Maddux BA, Hessler D, Goldfine ID, Youngren JF. Chromium supplementation in non-obese non-diabetic subjects is associated with a decline in insulin sensitivity. BMC Endocr Disord. 2012 Nov 30;12:31. doi: 10.1186/1472-6823-12-31. PMID 23194380